CLINICAL TRIAL: NCT02168556
Title: Interventions to Decrease Anxiety in Patients Undergoing Urodynamic Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-1351
Record Dates: First submitted 2014-05-27; First posted 2014-06-20 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Incontinence
Keywords: Urodynamics, Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy; Videotape Recording; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard of Care (Placebo Comparator): Patient underwent urodynamic testing by receiving only standard of care with mailed information and during test teaching.
  Interventions: Other: Standard of care
- Music (Active Comparator): Patient underwent urodynamic testing while listening to music that was 60 beats per minute and received standard of care information and teaching.
  Interventions: Behavioral: Music
- Video (Active Comparator): Patient watched an informational video prior to urodynamic testing.
  Interventions: Behavioral: Video

INTERVENTIONS:
Behavioral: Music — Subject listens to music that is 60bpm while undergoing urodynamic testing.
  Other Names: Music Therapy
  Arms: Music
Behavioral: Video — Subject watches an informational video prior to undergoing urodynamic testing.
  Other Names: Video therapy
  Arms: Video
Other: Standard of care — Standard of care
  Arms: Standard of Care

SUMMARY:
This is a randomized controlled trial to determine if music, a video, or standard of care will decrease anxiety in patients undergoing urodynamic testing.

DETAILED DESCRIPTION:
Research Design and Methods

This study was a randomized controlled trial assessing the interventions of music, a patient educational video, or usual care pre-test teaching practice and anxiety before patients undergo urodynamic testing. This study enrolled women who were scheduled to undergo urodynamic testing within the Female Pelvic Medicine and Reconstructive Surgery clinic on main campus and at Fairview Hospital. Consenting participants were randomized to receive either usual practice pre-test teaching, usual practice pre-test teaching with soothing music in the background and throughout the test, or usual practice pre-test teaching and watching an educational video before the test was performed. The participants filled out a short questionnaire before urodynamic testing was started with two VAS scales assessing anxiety and pain and Likert Scale Questions, a second short questionnaire when the patient feels "strong urge" with two VAS scales assessing anxiety and pain, and a third questionnaire once the patient has completed the test again testing VAS anxiety and pain as well as some Likert scale questions.

The primary outcome was to determine if pre-urodynamic testing anxiety was decreased after watching a pre-test educational video, or by listening to music before and throughout the procedure, or by receiving standard of care pre-test teaching. Secondary outcomes were to determine baseline anxiety in our urodynamic patient population and to determine if there is decreased discomfort due to the intervention as well as to evaluate if there were certain patients that would benefit from increased information.

Enrollment All patients undergoing urodynamic testing for the first time who are over the age of 18 years old, female with presentation for urodynamics for urinary dysfunction, urinary incontinence, prolapse, or presurgical evaluation of voiding function were screened for participation in the study.

Exclusion criteria included:

1. Pregnancy
2. Ongoing infections
3. Inability to cooperate
4. Inability to give consent
5. Non-English speakers
6. Patients who had undergone urodynamic testing in the past

Randomization

Random treatment assignments were placed in advance in set of sealed envelopes by a person who was not involved in opening the envelopes. Each envelope was numbered. When a patient was randomized, the patients name and the number of the next unopened envelope were recorded in a secure database. The envelope was then pened and the randomization was determined for the patient.

Data Collection Protocol

This study was incorporated into the patient's routine urodynamic testing. No additional visits were necessary.

Demographic data including patient's age, ethnicity, education, catheter history, mental health history and medications were obtained, and patient satisfaction with care scores were also be collected. Paper forms will be stored in the locked research office at the Cleveland Clinic. Questionnaires were then collected in REDcap, a secure, web-based application designned to support data capture. We de-identified each patient and did not include their name or Cleveland Clinic medical record number on our data collection sheet form or on the questionnaires, or in the database. During abstraction, a separate log was kept with patient identifying information and linking it to the database in case it was necessary to go back to the medical record to clarify or complete data entry. This log will be destroyed after data collection is complete and before data analysis. The database was kept on a password protected Gynecology research drive accessible only by the study investigators.

1. Patients randomized to the usual care arm woul have received mailings about urodynamic testing prior to arriving to the urodynamic suite. They then entered the urodynamic suite and the urodynamics provider discussed the information that was mailed to them. They also discussed the overall test, placement of catheters, and filling of the bladder with the patient before the provider began the test which is usual care. Once the provider finished giving the information, the patient filled out the first pre-test questionnaire which involved multiple Likert scale questions as well as Visual Analog Scale questions. During the urodynamic testing when the patient reached the point of "strong urge," a two question visual analog scale was given to the patient measuring anxiety and discomfort. Once the test has been concluded, the patient was given one further short post-test questionnaire using the Likert scale and Visual Analog Scale.
2. Patients randomized to the video arm arrived to their appointment having received the mailed material (usual practice). Prior to watching the video, the patient was given the pre-test questionnaire. While in the urodynamics suite the patient watched a short patient informational video on urodynamics. Urodynamic testing was then performed and when the patient noted "strong urge"during the testing period, a short, two question visual analog scale questionnaire measuring anxiety and discomfort was given. Once the urodynamic testing was completed, the patient will fill out an additional Likert scale and Visual Analog Scale post-test questionnaire.
3. Patients randomized to the music arm arrived to the appointment after having received mailed information about the test. The patient enter the urodynamics suite, was randomized and then slow music (tempo of 60 beats min) was started to play in the background. Usual practice instructions were given. The music continued through the urodynamic testing. Before the test and the usual practice instructions were given, the patient was given the pre-test questionnaire. When the patient notified the test provider that she had "strong urge" a second questionnaire with visual analog scales measuring anxiety and discomfort were given. Once the urodynamic testing was concluded, the patient was given the post-test questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above,
* female
* urinary dysfunction
* urinary incontinence
* prolapse
* presurgical evaluation of voiding function
* Never undergone Urodynamics before

Exclusion Criteria:

* Pregnancy
* Ongoing urinary tract infections
* Inability to cooperate
* Inability to give consent
* Non-English speakers
* Patients who have undergone urodynamic testing in the past

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Anxiety | One day
  The primary outcome is to determine if pre-urodynamic testing anxiety is decreased after watching a pre-test educational video, or by listening to music before and throughout the procedure, or by receiving standard of care pre-test teaching. For measurement of anxiety we used 100mm Visual analog scales. We used a questionnaire to obtain demographics. We used a five point Likert scale to ask questions about their use of the internet and information seeking behavior.

SECONDARY OUTCOMES:
Discomfort | One Day
  Secondary outcomes are to determine baseline anxiety in our urodynamic patient population and to determine if there is decreased discomfort due to the intervention as well as to evaluate if there are certain patients that would benefit from increased information. For measurement of discomfort we used 100mm Visual analog scales. We used a questionnaire to obtain demographics. We used a five point Likert scale to ask questions about their use of the internet and information seeking behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen R Solomon, MD, Principal Investigator — The Cleveland Clinic; Beri Ridgeway, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio

REFERENCES:
- [Derived] Solomon ER, Ridgeway B. Interventions to decrease pain and anxiety in patients undergoing urodynamic testing: A randomized controlled trial. Neurourol Urodyn. 2016 Nov;35(8):975-979. doi: 10.1002/nau.22840. Epub 2015 Jul 30. PMID 26227401